CLINICAL TRIAL: NCT03144765
Title: Multicenter Phase II Study of Transanal Total Mesorectal Excision (taTME) With Laparoscopic Assistance for Rectal Cancer
Brief Title: Multicenter Phase II Study of Transanal TME (taTME)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Society of American Gastrointestinal and Endoscopic Surgeons (Other); Research Foundation of the American Society of Colon and Rectal Surgeons (Other)
Responsible Party: Principal Investigator, Patricia Sylla, Associate Professor, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 16-2009
Record Dates: First submitted 2017-05-05; First posted 2017-05-09 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Rectal Cancer; Surgery
Keywords: taTME; Transanal; Rectal cancer; Colorectal; Total mesorectal excision; TME
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- taTME (Experimental): Enrolled subjects will undergo the study procedure, laparoscopically-assisted Transanal Total Mesorectal Excision (taTME).
  Interventions: Procedure: Transanal Total Mesorectal Excision (taTME)

INTERVENTIONS:
Procedure: Transanal Total Mesorectal Excision (taTME) — Study procedures consist in 1-team (sequential) or 2-team (combined) low anterior resection with transanal TME using laparoscopic or robotic abdominal assistance.
  Other Names: taTME

SUMMARY:
Radical rectal cancer resection, namely total mesorectal excision (TME), is the cornerstone of the treatment of resectable rectal cancer. In combination with chemotherapy and radiation treatment (CRT), complete TME with negative resection margins is associated with sustained local and systemic control even in locally advanced disease. Over the last 2 decades, laparoscopic and robotic techniques have been increasingly adopted due to reduced surgical trauma and faster patient recovery. Yet, both approaches are associated with equivalent postoperative morbidity and disturbances in sexual, urinary and defecatory function relative to open TME. Furthermore, laparoscopic and robotic TME remain associated with substantial conversion rates and variable rates of TME completeness as a result of the procedural difficulties reaching the low rectum from the abdominal approach. Transanal TME (taTME) with laparoscopic assistance was developed to facilitate completion of TME using a primary transanal endoscopic approach. Transanal TME uses a "bottom-up approach" to overcome the technical difficulties of low pelvic dissection using an abdominal approach. Published results from single-center taTME series and an international registry suggest the short-term procedural and oncologic safety of this approach in resectable rectal cancer. No multicenter phase II study has yet been conducted to validate the procedural safety, functional outcomes or long-term oncologic outcomes of this approach.

Study Design: This is a 5-year phase II multicenter single-arm study to evaluate the safety and efficacy of low anterior resection (LAR) with taTME using laparoscopic or robotic assistance in 100 eligible subjects with resectable rectal cancer.

Hypothesis: taTME is non-inferior to standard LAR with respect to the quality of the TME achieved.

DETAILED DESCRIPTION:
The management of rectal cancer is multidisciplinary and outcomes are dependent on accurate preoperative staging, performance of a curative resection, and the selective use of neoadjuvant and adjuvant therapy to improve long-term oncologic outcomes. Despite the increasing use of laparoscopic and robotic approaches, radical rectal cancer resection is associated with relatively high rates of conversion to open surgery, variable rates of TME specimen completeness, and morbidity rates that are equivalent to that of open TME with respect to infectious and wound-related complications, as well as defecatory, sexual and urinary dysfunction,.

Transanal TME (taTME) with laparoscopic assistance was developed in an effort to facilitate completion of TME using a primarily transanal endoscopic approach. Based on the preliminary results from several published single-center case series and the first international taTME registry, in carefully selected patients with resectable rectal cancer, taTME with laparoscopic assistance is associated with perioperative outcomes and short-term oncologic outcomes that are equivalent to that of standard TME.

This study is the first phase II multicenter trial of taTME conducted in the United States to evaluate the efficacy and safety of taTME with laparoscopic or robotic assistance relative to standard LAR. A total of 100 subjects with resectable rectal cancer located up to 10 cm from the anal verge will be enrolled across 10 US study sites. It is anticipated that this larger, phase II multicenter study will validate the safety and efficacy of taTME with respect to perioperative outcomes, short and long-term oncologic outcomes and functional results.

Study procedure:

Study procedures will consist in 1-team (sequential) or 2-team (combined) LAR with transanal TME using laparoscopic or robotic abdominal assistance. Laparoscopic or robotic abdominal access will be obtained followed by inferior mesenteric vessels transection, mobilization or the proximal colon and splenic flexure takedown if indicated. Transanal TME is performed either at the same time or following the above steps. Intersphincteric resection (ISR) may be included for very low tumors. Following pursestring closure of the rectum below the tumor, transanal endoscopic TME dissection will proceed circumferentially until the peritoneal cavity is entered anteriorly. Following complete mobilization of the rectosigmoid, the specimen is extracted transanally or transabdominally followed by colorectal or coloanal anastomosis, with or without a diverting loop ileostomy. Operative details will be recorded in case report forms (CRF's).

TME pathology assessment:

Resected specimens will be processed and analyzed by the participating institution's Pathology Department according to standard TME protocol. De-identified photographs of all fresh TME specimens will be independently reviewed by a Pathology Review Committee blinded to the source of the specimen.

Postoperative care and follow-up:

Subjects will be managed according to standard postoperative protocols. Postoperative visits and oncology follow-up visits will occur as per standard practice and oncologic outcomes. All adverse events occurring during the study period will be graded using the Clavien-Dindo system. Postoperative functional questionnaires will be obtained 6-8 months and 12-14 months postoperatively in non-diverted subjects. In diverted subjects, functional questionnaires will be collected 3-4 months and 9-10 months following ileostomy closure (or 12-18 months following the study procedure).

ELIGIBILITY:
Inclusion Criteria:

* New diagnosis of histologically confirmed adenocarcinoma of the rectum
* Age ≥18
* Clinical stage cT1 (high-risk), T2, or T3, cN0, N1, N2 on staging pelvic MRI
* Negative predicted CRM on staging pelvic MRI
* No evidence of metastasis on CT scans of the chest, abdomen and pelvis
* Rectal cancer located within 10 cm from the anal verge based on proctoscopy and digital rectal examination (DRE)
* Complete preoperative colonoscopy demonstrating no synchronous colon cancer
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 (Karnofsky ≥ 60%)
* Eligible to undergo laparoscopic or robotic LAR with or without a temporary diverting stoma, based on multidisciplinary tumor board consensus
* Able to understand and willing to sign a written informed consent form

Exclusion Criteria:

* cT4 on staging pelvic MRI
* >12 weeks delay between completion of neoadjuvant CRT and planned study procedure
* Severely symptomatic rectal tumors
* Tumors invading into the internal anal sphincter muscle based on DRE and pelvic MRI
* Fecal incontinence at baseline
* Prior history of rectal resection
* Prior history of colorectal cancer
* History of inflammatory bowel disease
* Uncontrolled concurrent illness
* Pregnancy
* Subjects who cannot read or understand English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-09-25 (Actual); Primary Completion 2022-04-12 (Actual); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Quality of Mesorectal Excision | 30 days
  Rate of complete and near-complete mesorectal excision achieved with taTME, based on standard pathologic assessment of TME specimens.

SECONDARY OUTCOMES:
Complete pathology assessment of TME specimens | 30 days
  TNM grading, margins assessment
30-day perioperative complications | 30 days
  The rate of complications experienced intraoperatively and postoperatively (within 30 days of the study procedure)
Long-term postoperative complications | 12 months
  Incidence of long-term term postoperative complications
Change in COREFO scores | 18 months
  Alterations in Colorectal Functional Outcome Questionnaire (COREFO) scores from baseline up to 18 months postoperatively - 27 items. All questions can be answered by choosing from five response options; No; Never; Yes, less than once a week; Yes, 1-2 days per week; Yes, 3-5 days per week; Yes, 6-7 days per week.
Change in FIQLscores | 18 months
  Alterations in Fecal Incontinence Quality of Life Instrument (FIQL) scores from baseline up to 18 months postoperatively - 29 items range from 1 (strongly agree) to 4 (strongly disagree); with a 1 indicating a lower functional status of quality of life. Scale scores are only calculated if at least half of the items have been answered.
Change in Wexner score | 18 months
  Alterations in Wexner score from baseline up to 18 months postoperatively. Wexner questionnaire - 5 questions and scored from 0 = never to 4= always, with total score from 0 (no incontinence) to 20 (complete incontinence)
Change in International Index of Erectile Function [IIEF] score | 18 months
  Alterations in IIEF scores from baseline up to 18 months postoperatively - 15 item questionnaire, each item range from 0 - 5, with total score to 30. lower score indicates more severe erectile dysfunction (ED)
Change in Female Sexual Function Index [FSFI] | 18 months
  Alterations in FSFI from baseline up to 18 months postoperatively - 19-item self-report measure, each item ranges from 0-5, with full range from 2 to 36, with low score indicating sexual function disorder.
Change in IPSS | 18 months
  Alterations in International Prostate Symptom Score (IPSS) from baseline up to 18 months postoperatively - IPSS 8 questions total - 7 questions related to symptoms, each item scored 1-5. (asymptomatic to very symptomatic). The 8th question refers to the patient's perceived quality of life ranged from 0 to 6 ("delighted" to "terrible".) Total scale ranges from 8-35. Mild (symptom score less than of equal to 7), Moderate (symptom score range 8-19), Severe (symptom score range 20-35).
3-year oncologic outcomes | 3-5 years
  3-year local recurrence rate, distant recurrence rate, disease-free survival and overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Sylla, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (12):
- United States (11):
  - Kaiser Permanente, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - UC Irvine Hospital, Orange, California
  - Florida Hospital, Orlando, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - University of Massachusetts, Worcester, Massachusetts
  - Mount Sinai Beth Israel, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Providence Portland Medical Center, Portland, Oregon
  - Lankenau Institute, Wynnewood, Pennsylvania
- Toronto Western Hospital, Toronto, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sylla P, Sands D, Ricardo A, Bonaccorso A, Polydorides A, Berho M, Marks J, Maykel J, Alavi K, Zaghiyan K, Whiteford M, Mclemore E, Chadi S, Shawki SF, Steele S, Pigazzi A, Albert M, DeBeche-Adams T, Moshier E, Wexner SD. Multicenter phase II trial of transanal total mesorectal excision for rectal cancer: preliminary results. Surg Endosc. 2023 Dec;37(12):9483-9508. doi: 10.1007/s00464-023-10266-9. Epub 2023 Sep 12. PMID 37700015
- See also: Study description on SAGES website — https://www.sages.org/tatme-study/

DOCUMENTS (1):
  • Informed Consent Form (2021-09-13): https://cdn.clinicaltrials.gov/large-docs/65/NCT03144765/ICF_000.pdf